CLINICAL TRIAL: NCT01722344
Title: Individual Placement and Support (IPS) Enhanced With Cognitive Remediation and Social Skills Training in Denmark: a Randomized Controlled Trial
Brief Title: Improving Work Outcome for People With Severe Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Odense University Hospital (Other); Copenhagen Municipality, Denmark (Other Government); Odense Municipality (Unknown); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Silkeborg Municipality (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PCK-2012-CT-2912
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Schizophrenia, Schizotypal and Delusional Disorders; Bipolar Affective Disorder; Recurrent Depressive Disorder
Keywords: Severe mental illness; Vocational rehabilitation; Supported employment; Individual placement and support; Cognitive remediation; Social skill training
MeSH Terms: conditions — Schizophrenia; Schizophrenia, Paranoid; Bipolar Disorder; Depressive Disorder; Mental Disorders | interventions — Palliative Care; Myo-Inositol-1-Phosphate Synthase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Individual Placement and Support (IPS) (Experimental)
  Interventions: Behavioral: Individual Placement and support (IPS)
- IPS plus (Experimental): Individual Placement and Support plus cognitive remediation and work-related social skills training
  Interventions: Behavioral: Individual Placement and support (IPS); Behavioral: IPS plus
- Standard intervention (No Intervention)

INTERVENTIONS:
Behavioral: Individual Placement and support (IPS) — IPS involves an employment specialist who is integrated within the mental health team, and carries out all phases of the vocational services, with a caseload on less than 25. The intervention is based on the 7 principles of IPS Supported Employment. The essence of these principles is an individualized and rapid search for competitive employment or education that avoids prolonged prevocational training and preparation. The intervention is integrated within the mental health services, with emphasis on client preference and choice regarding jobs, and with availability of on going job support and benefit counselling
  Arms: IPS plus; Individual Placement and Support (IPS)
Behavioral: IPS plus — Individual Placement and Support + cognitive remediation and work-related social skills training, consists of the IPS intervention + 24 sessions of computer based cognitive training and 24 group based sessions of cognitive coping strategies and work-related social skills training.
  Arms: IPS plus

SUMMARY:
The purpose of this study is to investigate the efficacy of IPS in Denmark and compare effects of 1. Individual Placement and Support (IPS) vs. 2. IPS + cognitive remediation and work-related social skills training vs. 3. standard intervention, among individuals with severe mental illness.

DETAILED DESCRIPTION:
Individual Placement and Support (IPS) is established as the most effective vocational intervention available for persons with severe mental illness,and the intervention is widely recognized as an evidence-based practice. Despite evidence, long-term job retention and economic self-sufficiency have not been clearly demonstrated. Research has suggested that integrating methods such as cognitive remediation and social skills training could reduce such limitations. Further, there has not been conducted any randomized controled trials with IPS in Scandinavian countries with highly developed and generous social security and welfare systems, and with high thresholds to the open labour market.

The aim of this study is to investigate the effectiveness of IPS in Denmark and compare effects of 1. IPS vs. 2. IPS + cognitive remediation and work-related social skills training vs. 3. Standard intervention.

The intervention is based on the 7 principles of IPS Supported Employment, and IPS enhanced with cognitive remediation and work-related social skills training, consists of 24 sessions of computer based cognitive training and 24 group based sessions of cognitive coping strategies and work-related social skills training.

ELIGIBILITY:
Inclusion Criteria:

Psychosis within the schizophrenic spectrum (F 2, International Classification of Diseases (ICD 10)).

Severe depression (F33, ICD-10) or Bipolar disorder (F31, ICD-10) and minimum 3 years psychiatric treatment.

Motivated for employment or education. 18 to 65 years old. Participants must speak and understand Danish.

Exclusion Criteria:

Lack of informed consent Above 64 years and receiving state pension Match group 1 (No problems besides unemployment)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 717 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Hours in competitive employment or education | Measured at 18 month

SECONDARY OUTCOMES:
In competitive employment or education at some point during follow up period | Measured at 18 month follow-up
Days to first employment or beginning of education | Measured at 18 month follow-up
Average monthly earnings in follow-up period | Measured at 18 month follow-up
Hours of work per week among those who obtain competitive employment during the follow-up period | Measured at 18 month follow-up
Negative symptoms measured with Schedule for assessment of negative symptoms in schizophrenia (SANS) | Measured at 18 month follow-up
Cognitive functions measured with The Brief Assessment of Cognition in Schizophrenia (BAC) | Measured at 18 month follow-up
Functioning measured with Global Assessment of Functioning (GAF) | Measured at 18 month follow-up
Functioning measured with Personal and Social Performance (PSP) | Measured at 18 month follow-up
Quality of life measured with SF-12 | Measured at 18 month follow-up
Empowerment measured with Empowerment Scale | Measured at 18 month follow-up
Self-efficacy measured with General self-efficacy scale (GSE) | Measured at 18 month follow-up
Self-esteem measured with The Rosenberg Self-Esteem scale | Measured at 18 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Eplov, MD, Phd, Study Director — Copenhagen University Hospital, Mental Health Centre Copenhagen; Merete Nordentoft, Professor, Principal Investigator — Copenhagen University Hospital, Mental Health Centre Copenhagen; Elsebeth Stenager, MD, Phd, Principal Investigator — Department of Psychiatry, Odense, The University of Southern Denmark.; Bent Nielsen, Professor, Principal Investigator — Department of Psychiatry, Odense, The University of Southern Denmark
Locations (1):
- Mental Health Centre Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Christensen TN, Wallstrom IG, Stenager E, Bojesen AB, Gluud C, Nordentoft M, Eplov LF. Effects of Individual Placement and Support Supplemented With Cognitive Remediation and Work-Focused Social Skills Training for People With Severe Mental Illness: A Randomized Clinical Trial. JAMA Psychiatry. 2019 Dec 1;76(12):1232-1240. doi: 10.1001/jamapsychiatry.2019.2291. PMID 31483451
- [Derived] Christensen TN, Nielsen IG, Stenager E, Morthorst BR, Lindschou J, Nordentoft M, Eplov LF. Individual Placement and Support supplemented with cognitive remediation and work-related social skills training in Denmark: study protocol for a randomized controlled trial. Trials. 2015 Jun 21;16:280. doi: 10.1186/s13063-015-0792-0. PMID 26093636